CLINICAL TRIAL: NCT06421038
Title: Efficacy of Thyme Honey in The Management of Oral Aphthous Ulcers: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Thyme Honey in The Management of Oral Aphthous Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-031
Record Dates: First submitted 2024-05-07; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Aphthous Stomatitis (Major) (Minor); Treatment Compliance
Keywords: Oral diseases; Thyme honey; anti-inflammatory; natural products
MeSH Terms: conditions — Stomatitis, Aphthous; Patient Compliance | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Thyme honey on recurrent aphthous stomatitis
Who Masked: Care Provider, Outcomes Assessor
Masking Description: the care provider and the outcomes assessor will not know which treatment will be given to the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyme honey (Experimental): 10 patients will be treated by thyme honey application (100% pure natural honey, applied by themselves) on their ulcers three times a day for 7 days.
  Interventions: Other: Thyme honey
- kenalog in orabase (Active Comparator): 10 patients will be treated by kenalog in orabase (Triamcinolone acetonide 0.1% in oral paste 5g), three times a day for 7 days only.
  Interventions: Drug: Kenalog

INTERVENTIONS:
Other: Thyme honey — Thyme honey is a rich monofloral honey variety formed by bees that collect nectar from thymus vulgaris flowers. thyme honey application (100% pure natural honey, applied by themselves) on their ulcers three times a day for 7 days
  Arms: Thyme honey
Drug: Kenalog — kenalog in orabase (Triamcinolone acetonide 0.1% in oral paste 5g)
  Other Names: kenalog in orabase
  Arms: kenalog in orabase

SUMMARY:
Recurrent aphthous stomatitis (RAS) is considered the most common oral mucosal lesion, present first in childhood or adolescence. Aphthous ulcers affect up to 25% of the general population, and 3-month recurrence rates are as high as 50%, it is more common in female, also it increases by increasing age and minor aphthous ulcers are 80% of suffered patient.

Due to the antimicrobial, anti-inflammatory, antifungal, and analgesic effects of Thyme honey, and the lack of evidence in the considered population, the present study aimed to assess the effect of honey on the pain relief in patients with minor RAU as a primary objective and to assess the healing effect of natural thyme honey on minor RAU, and the Oral Health Impact Profile (OHIP-14) as a secondary objectives.

DETAILED DESCRIPTION:
Treatment of aphthous will usually be for three purposes: reduction of pain and inflammation, prevention of secondary infection, reduction of duration and repetition of aphthous. The most common treatments, after oral hygiene, are: use of local and oral steroids that have effect on T-lymphocytes and reduce inflammation, use of local antibiotics, for example, chlorohexidine, benzidamine, solving vitamin and mineral deficiency, such as B12, iron, folic acid, and avoidance of food allergens. Other treatments such as amelexanox, a potent inhibitor of inflammation due to mast cells and neutrophils. levamisol, talidomide are effective too.

Many factors may be involved in its progression, such as genetic predisposition, immunological abnormalities, microbial infection, psychological stress, and hormonal state. Since the etiology and pathogenesis of RAS remains unclear, there is currently no consensus regarding a definitive curative therapy. The commonly accepted treatment strategy is to lessen the pain and duration of lesions. Topical corticosteroids, antibiotics, and analgesics are highly recommended for patients with RAS.

However, longer treatment and frequent exposure to these medications may cause fungal infection and drug resistance, which may further lead to more severe adverse effects or even life-threatening complications. Natural herbal medicines as an alternative therapy for RAS have been widely used in many countries for decade. Clinical studies on the use of such remedies have reported favorable benefits to patients by reducing the discomfort and duration of ulcers.

The large volume of literatures reported the effectiveness of honey. It indicates that it may potentially be useful to treat periodontal diseases, mouth ulcers and other problems of oral health. Furthermore, the application of honey to a wound has been demonstrated to stimulate the production and release of pro-inflammatory cytokines that assist in the wound healing process, such as interleukin-1 and tumor necrosis factor-alpha. The topical application of honey to various injured tissues has also been shown to stimulate wound repair through the stimulation of growth of epithelial cells, reduction of edema, and wound debridement.

Takzaree et al in 2017 have evaluated the effects of local application of thyme honey in open cutaneous wound healing and concluded that local application of honey two times per day could boost the healing process as it reduces the inflammation, increases granulation tissue formation, and promotes angiogenesis and epithelialization, and this would eventually result in a quicker wound healing process. These antioxidants and wound healing effects have also been validated for Tulkarm honey and Thymus vulgaris honey. A recent study revealed substantial beneficial effects of Thymus vulgaris honey on skin wound healing and recommended its use in various types of wounds.

Recent research aimed to evaluate the effect of thyme honey oral gel in the prevention of chemotherapy-induced oral mucositis in patients with breast cancer with an emphasis on patient-reported symptoms. The study concluded that the use of thyme honey oral gel reduced the incidence, duration, and severity of symptoms of oral mucositis, in addition to delaying the occurrence of grade ≥2 oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* • The study involved patients who had a positive history of having similar oral mucosal ulcers for 3-4 months and ulcers for <48 h.

  * Clinically diagnosed patients with chronic aphthous stomatitis measuring ≤5 mm in size in the oral cavity and who gave written consent for participation.
  * Only single ulcers were considered for the study.
  * Systemically health patients.

Exclusion Criteria:

* The study excluded patients with a history of associated systemic disease.

  * Cases of chronic aphthous stomatitis (major), lesions of herpetic form, numerous RAS lesions, and smoking.
  * In addition, no consideration was given to patients with a history of hypersensitivity to honey.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 7 days.
  Visual Analog Scale (0-10) will be used to determine the intensity of pain on day 0, day 3, day 5, and day 7.

SECONDARY OUTCOMES:
Size of ulcers (in mm) | 7 days.
  after starting treatment, ulcer size will be recorded on day 0, day 3, day 5, and day 7, using a calibrated dental probe with millimeter marking.
The Oral Health Impact Profile (OHIP-14) questionnaire | 7 days
  The Oral Health Impact Profile (OHIP-14) questionnaire has been assessed 1 week after intervention. OHIP-14 utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often). A lower score in any of the five categories indicates higher satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Confidentiality of data: All data will be stored in an Excel sheet for research purposes and respecting patient confidentiality. Patients have the right to withdraw from the research at any point for any reason and with no penalty subject to them.

REFERENCES:
- [Background] Bang LM, Buntting C, Molan P. The effect of dilution on the rate of hydrogen peroxide production in honey and its implications for wound healing. J Altern Complement Med. 2003 Apr;9(2):267-73. doi: 10.1089/10755530360623383. PMID 12804080
- [Background] Eisen D, Carrozzo M, Bagan Sebastian JV, Thongprasom K. Number V Oral lichen planus: clinical features and management. Oral Dis. 2005 Nov;11(6):338-49. doi: 10.1111/j.1601-0825.2005.01142.x. PMID 16269024
- [Background] Embil JA, Stephens RG, Manuel FR. Prevalence of recurrent herpes labialis and aphthous ulcers among young adults on six continents. Can Med Assoc J. 1975 Oct 4;113(7):627-30. PMID 1181018